CLINICAL TRIAL: NCT00550355
Title: A Randomized, Subject and Investigator-Blind, Placebo-Controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Intravenously Administered Doses of PD-0360324 in Patients With Rheumatoid Arthritis Receiving Methotrexate
Brief Title: Dose-Escalating Multiple Dose Study of PD-0360324 in Combination With Methotrexate in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6261002
Record Dates: First submitted 2007-10-25; First posted 2007-10-29 (Estimated); Last update posted 2009-07-14 (Estimated); Status verified 2009-07

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: PD 0360324
- 2 (Experimental)
  Interventions: Drug: PD 0360324
- 3 (Experimental)
  Interventions: Drug: PD 0360324
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PD 0360324 — 3 doses of PD 0360324 (Dose level 1) administered over 12 weeks
  Arms: 1
Drug: PD 0360324 — 3 doses of PD 0360324 (Dose level 2) administered over 12 weeks
  Arms: 2
Drug: PD 0360324 — 3 doses of PD 0360324 (Dose level 3) administered over 12 weeks
  Arms: 3
Drug: Placebo — 3 doses of Placebo administered over 12 weeks
  Arms: 4

SUMMARY:
This study is designed to evaluate the safety and tolerability of multiple intravenously administered doses of PD 0360324 in patients with rheumatoid arthritis receiving methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA for at least 6 months based upon the American College of Rheumatology (ACR) 1987 Revised Criteria.
* Must have been treated with methotrexate (≥7.5 mg/week to ≤25 mg/week) for at least 16 weeks immediately prior to enrollment. The dose of methotrexate must be stable for at least 6 weeks prior to enrollment.
* Females of childbearing potential are required to simultaneously use 2 effective contraceptive methods, 1 of which must be a barrier (condoms, diaphragm or cervical cap) with spermicide. Non-vasectomized men must be willing to abstain from sexual intercourse or willing to use a condom in addition to having their female partner use another form of contraception, if the woman could become pregnant from the time of the first dose of study medication until completion of follow up procedures
* Contact your local site for more inclusion criteria.

Exclusion Criteria:

* Diagnosis of any other inflammatory arthritis (eg, spondyloarthropathies); or a non-inflammatory arthritis or musculoskeletal condition (eg, osteoarthritis, fibromyalgia) that, in the investigator's opinion, may interfere with clinical assessments.
* Evidence of active or latent infection with Mycobacterium tuberculosis (TB).
* Use of etanercept, anakinra, or oral DMARDs with the exception of methotrexate, within the 4 weeks prior to enrollment. Use of biological DMARDs within the 8 (adalimumab or infliximab) or 12 (abatacept) or 56 (rituximab) weeks prior to enrollment. Use of oral corticosteroids, acetaminophen, NSAIDs, and opioids are permitted within the dose ranges defined in the protocol.
* Contact your local site for more inclusion criteria.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2007-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Clinical safety laboratories | 16 weeks
Vital signs | 16 weeks
ECG | 16 weeks
Incidence and severity of adverse events | 16 weeks

SECONDARY OUTCOMES:
Pharmacokinetic | 16 weeks
Pharmacodynamic | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (21):
- United States (8):
  - Pfizer Investigational Site, Peoria, Arizona
  - Pfizer Investigational Site, Daytona Beach, Florida
  - Pfizer Investigational Site, Port Orange, Florida
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Frederick, Maryland
  - Pfizer Investigational Site, Lansing, Michigan
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Dallas, Texas
- Pfizer Investigational Site, Buenos Aires, Argentina
- Bulgaria (2):
  - Pfizer Investigational Site, Pleven
  - Pfizer Investigational Site, Sofia
- Czechia (2):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Prague
- Mexico (2):
  - Pfizer Investigational Site, México, D.F.
  - Pfizer Investigational Site, Mexico City, Mexico City
- Poland (4):
  - Pfizer Investigational Site, Bialystok
  - Pfizer Investigational Site, Krakow
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Wroclaw
- Pfizer Investigational Site, Piešťany, Slovakia
- Pfizer Investigational Site, Santiago de Compostela, A CORUÑA, Spain

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6261002&StudyName=Dose-Escalating%20Multiple%20Dose%20Study%20of%20PD-0360324%20in%20Combination%20with%20Methotrexate%20in%20Patients%20with%20Rheumatoid%20Arthritis